CLINICAL TRIAL: NCT01937767
Title: A Randomized, Single-blind Phase II Study Evaluating the Efficacy, Safety and Pharmacokinetics of Remimazolam in General Anesthesia in Adult Patients Undergoing Cardiac Surgery, Including Follow-up Sedation in the PACU/ICU
Brief Title: Remimazolam Phase II Cardiac Anesthesia Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: Aptiv Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNS7056-010; 2013-001113-32 (EudraCT Number)
Record Dates: First submitted 2013-08-29; First posted 2013-09-10 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: General Anesthesia
MeSH Terms: interventions — remimazolam; Propofol; Sevoflurane; Remifentanil; WW Domain-Containing Oxidoreductase; Fentanyl; Rocuronium; Solutions; Injections

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propofol (Active Comparator): Induction: Propofol, fentanyl, rocuronium. Maintenance: Sevoflurane, remifentanil.
  Interventions: Drug: Propofol; Drug: Sevoflurane; Drug: Remifentanil; Drug: Fentanyl; Drug: Rocuronium
- Remimazolam 6 mg/kg/hr (Experimental): Induction: Remimazolam 6 mg/kg/hr, fentanyl, rocuronium. Maintenance: Remimazolam up to 2 mg/kg/hr titrated to effect, remifentanil.
  Interventions: Drug: Remimazolam; Drug: Remifentanil; Drug: Fentanyl; Drug: Rocuronium
- Remimazolam 12 mg/kg/hr (Experimental): Induction: Remimazolam 12 mg/kg/hr, fentanyl, rocuronium. Maintenance: Remimazolam up to 2 mg/kg/hr titrated to effect, remifentanil.
  Interventions: Drug: Remimazolam; Drug: Remifentanil; Drug: Fentanyl; Drug: Rocuronium

INTERVENTIONS:
Drug: Remimazolam
  Other Names: ByFavo, Aptimyda, CNS7056
  Arms: Remimazolam 12 mg/kg/hr; Remimazolam 6 mg/kg/hr
Drug: Propofol
  Other Names: Propofol-®Lipuro 10 mg/ml
  Arms: Propofol
Drug: Sevoflurane
  Other Names: Sevofluran Baxter
  Arms: Propofol
Drug: Remifentanil
  Other Names: Ultiva (remifentanil hydrochloride) for Injection
Drug: Fentanyl
  Other Names: Fentanyl-Janssen
Drug: Rocuronium
  Other Names: Esmeron 10mg/ml solution for injection

SUMMARY:
This phase II study in patients undergoing elective cardiac surgery will evaluate the efficacy, safety, and pharmacokinetics of remimazolam, compared with propofol and sevoflurane, during the induction and maintenance of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for major elective cardiac surgery.
* scheduled for mechanical ventilation via tracheal intubation.

Exclusion Criteria:

* thoraco-abdominal replacement of the aorta or other procedure expected to be accompanied by a massive hemorrhage (at least 15% of the circulating blood volume).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with successful anesthesia | Between the start of study medication and the end of the surgical procedure (up to approx 12 hours)
  Successful anesthesia was defined as no use of rescue sedative medication between start of the study medication and end of the surgical procedure completion of last skin suture.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Probst, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- Herzzentrum Leipzig GmbH, Leipzig, Germany